CLINICAL TRIAL: NCT03442257
Title: PUSH ME (Primary Care USage of Health Promoting Messages): A Text Message-based Intervention for Prevention of Cardiovascular Disease in Primary Care Patients With Hypertension: a Randomized Controlled Pilot Trial
Brief Title: Text Message Intervention for Prevention of Cardiovascular Disease in Primary Care Patients With Hypertension
Acronym: PUSH-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/674
Record Dates: First submitted 2018-01-11; First posted 2018-02-22 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-02

CONDITIONS: Hypertension; Cardiovascular Risk Factor
Keywords: Hypertension; Text Messaging; Primary Prevention; Cardiovascular Risk Factor; Primary Health Care; Health Promotion
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The research assistant, the patients' GPs, as well as all researchers except one (MS) will be blinded to group allocation. If the patients have questions regarding the SMS function they will be able to contact MS for help.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMS group (Experimental): Participants in the intervention group will receive four semi-personalized messages per week in addition to their usual care according to the National Board of Health and Welfare guidelines for hypertension treatment.
  Interventions: Behavioral: SMS
- Control (No Intervention): The control group will receive usual care according to the National Board of Health and Welfare guidelines for hypertension treatment.

INTERVENTIONS:
Behavioral: SMS — The experimental treatment will consist of health promoting text messages addressing metabolic risk factors associated with cardiovascular disorders in patients with hypertension. Participants will receive four semi-personalized messages per week in addition to their usual care. The text messages will be developed to support healthy life style changes i.e. regarding general cardiovascular health, tobacco use, physical activity and diet.
  Arms: SMS group

SUMMARY:
The primary objective of the study is to examine the impact of lifestyle advices, administered through regularly sent SMS, on hypertension in a primary health care setting. The secondary objective is to evaluate changes in other cardiovascular risk factors and general health, e.g. tobacco use, obesity, blood lipids, blood glucose, self-rated health and health-related quality of life.

DETAILED DESCRIPTION:
Background- The globalization of unhealthy lifestyles and demographic ageing of the world's population has contributed to the fact that high blood pressure is classified by World Health Organization as the world's leading risk for mortality.

Persistent hypertension is a key risk factor for coronary heart disease (CHD), stroke and other cardiovascular diseases (CVD), such as heart failure. CVD is, despite a decline in recent decades, still the leading cause of death in Sweden (4). The prevalence of hypertension in adults is around 40% according to a recent multinational study (5). In 30-40% of hypertensive individuals, additional metabolic risk factors such as dyslipidemia, insulin resistance and elevated glucose occur simultaneously, which further multiply the risk for heart disease, diabetes and stroke. An unhealthy lifestyle with physical inactivity and excess energy intake is the major driver of these metabolic risk factors. In most cases lifestyle intervention can reverse or reduce the unfavorable metabolic profile.

Primary healthcare in Sweden is managing the first-line healthcare, offering both prevention and treatment for a majority of chronic diseases. In Sweden, the vast majority of patients with hypertension are treated in primary health care. If the hypertension is well controlled, the GP typically meets the patient once a year for medical checkup, blood tests and medical prescription.

Interventions by SMS-texting have been shown to significantly improve compliance to medications, follow-up rate or disease monitoring.

Trial Design - Randomised clinical trial

Intervention - The experimental treatment will consist of an SMS-intervention addressing metabolic risk factors associated with cardiovascular disorders in patients with hypertension.

After baseline measurement participants in the intervention group will receive four semi-personalized messages per week in addition to their usual care according to the National Board of Health and Welfare guidelines for hypertension treatment. The text messages will be developed to support healthy life style changes i.e. regarding general cardiovascular health, tobacco use, physical activity and diet.

Control Treatment - The control group will receive usual care according to the National Board of Health and Welfare guidelines for hypertension treatment.

Recruitment - The participants will be recruited consecutively from three different PHCCs in Skåne. Patients with hypertension will receive information about the study at their annual check-up or other appointment with their GP. If they choose to participate, they will be contacted by phone by a research assistant for additional information, possibility to ask questions about the study, and scheduling a baseline control at their PHCC.

Baseline examination - Included patients that consent to take part in the study will be invited to their PHCC for a baseline visit. The following measurements will be assessed by a research assistant: blood pressure (in sitting position after 5 minutes rest; mean of two measurements in a standardized procedure with validated electronic BP devices), BMI and waist-hip circumference. Furthermore, the patients will complete a short questionnaire for evaluation of medical history, medication, tobacco and alcohol use, physical activity level, self-rated health and health-related quality of life. Blood samples for fasting plasma glucose, HbA1c and cholesterol will be drawn in the morning within a few days after the baseline visit.

Randomization- Randomization to study groups will be performed after completion of baseline assessments and questionnaires. A computer generated random number schedule with block sizes of four will be prepared. To assure allocation concealment, the information about group affiliation will be delivered through sealed envelopes.

The research assistant, the patients' GPs, as well as all researchers except Magnus Sandberg (MS) will be blinded to group allocation. If the patients have questions regarding the SMS function they will be able to contact MS for help.

Follow up- Follow up control will be performed after 6 months with the same assessments as at the baseline visit.

Power and sample size - For the pilot study we have assumed that a total number of 60 patients (20 patients per PHCC) will be sufficient to evaluate the feasibility of the intervention and the logistics of the assessments.

For the future full scale study, each group must contain 143 participants. The sample size is based on an assumed statistical power of 80 %, a two-sided test, a significance level of 5 %, a difference of 5 mm Hg between the groups, a standard deviation of 14 mm Hg and a drop out rate of 15 %.

Analysis plan - Data will be analysed according to the Intention-to-treat principle. Differences in mean change of end points between intervention and control groups will be calculated by ANCOVA, with baseline values as covariates.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hypertension (defined by the International classification of disease Manual ICD-10, diagnose code I10.9).
2. 40 to 80 years of age
3. Patient must own a mobile phone compatible with SMS

Exclusion Criteria:

1. History of myocardial infarction, stroke, transient ischemic attack (TIA), claudicatio intermittens, abdominal aortic aneurysm, previous heart surgery i.e. PCI or bypass (reported by recruiting physician or by patient in the questionnaire)
2. Blood pressure at baseline visit ≥180/110 mmHg or systolic blood pressure <120 mmHg.
3. Serious illness, other than cardiovascular, with short life expectancy (<1 year)
4. Predicted inability to comply with the study protocol e.g. language difficulties, interpreter needs, serious cognitive impairment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Six months
  Measured by automated devices (mmHg)

SECONDARY OUTCOMES:
Changes in cholesterol | six months
  Measured by blood test, total cholesterol (mmol/l)
Changes in high-density lipoprotein [HDL] | six months
  Measured by blood test, high-density lipoprotein [HDL] (mmol/l)
Changes in low-density lipoprotein [LDL] | six months
  Measured by blood test, low-density lipoprotein [LDL] (mmol/l)
Changes in tobacco use | six months
  Self-reported
Changes in BMI | six months
  Measured by research assistant at baseline and follow up (weight and hight will be combined to report BMI in kg/m2)
Changes in Blood glucose | six months
  HbA1c
Changes in self-rated health | six months
  five-graded Likert scale from excellent to poor. The question posed is; in general, would you say that you health is excellent, very good, good, fair, or poor?
Changes in self rated quality of life | six months
  EQ5D-5L (EuroQol 5 dimentions).The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'.
Changes in level of physical activity | six months
  self-reported physical activity
Changes in alcohol use | six months
  self-reported

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Lomma vårdcentral, Lomma, Skåne County
  - Löddeköpinge vårdcentral, Löddeköpinge, Skåne County
  - Sorgenfri vårdcentral, Malmo, Skåne County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in blood pressure from 1975 to 2015: a pooled analysis of 1479 population-based measurement studies with 19.1 million participants. Lancet. 2017 Jan 7;389(10064):37-55. doi: 10.1016/S0140-6736(16)31919-5. Epub 2016 Nov 16. PMID 27863813
- [Background] Chow CK, Teo KK, Rangarajan S, Islam S, Gupta R, Avezum A, Bahonar A, Chifamba J, Dagenais G, Diaz R, Kazmi K, Lanas F, Wei L, Lopez-Jaramillo P, Fanghong L, Ismail NH, Puoane T, Rosengren A, Szuba A, Temizhan A, Wielgosz A, Yusuf R, Yusufali A, McKee M, Liu L, Mony P, Yusuf S; PURE (Prospective Urban Rural Epidemiology) Study investigators. Prevalence, awareness, treatment, and control of hypertension in rural and urban communities in high-, middle-, and low-income countries. JAMA. 2013 Sep 4;310(9):959-68. doi: 10.1001/jama.2013.184182. PMID 24002282
- [Background] Schillaci G, Pirro M, Vaudo G, Gemelli F, Marchesi S, Porcellati C, Mannarino E. Prognostic value of the metabolic syndrome in essential hypertension. J Am Coll Cardiol. 2004 May 19;43(10):1817-22. doi: 10.1016/j.jacc.2003.12.049. PMID 15145106
- [Background] Grundy SM. Metabolic syndrome update. Trends Cardiovasc Med. 2016 May;26(4):364-73. doi: 10.1016/j.tcm.2015.10.004. Epub 2015 Oct 31. PMID 26654259
- [Background] Lin H, Wu X. Intervention strategies for improving patient adherence to follow-up in the era of mobile information technology: a systematic review and meta-analysis. PLoS One. 2014 Aug 6;9(8):e104266. doi: 10.1371/journal.pone.0104266. eCollection 2014. PMID 25100267
- [Background] Krishna S, Boren SA, Balas EA. Healthcare via cell phones: a systematic review. Telemed J E Health. 2009 Apr;15(3):231-40. doi: 10.1089/tmj.2008.0099. PMID 19382860
- [Background] Bengtsson U, Kjellgren K, Hallberg I, Lindwall M, Taft C. Improved Blood Pressure Control Using an Interactive Mobile Phone Support System. J Clin Hypertens (Greenwich). 2016 Feb;18(2):101-8. doi: 10.1111/jch.12682. Epub 2015 Oct 12. PMID 26456490
- [Background] Chow CK, Redfern J, Hillis GS, Thakkar J, Santo K, Hackett ML, Jan S, Graves N, de Keizer L, Barry T, Bompoint S, Stepien S, Whittaker R, Rodgers A, Thiagalingam A. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1255-63. doi: 10.1001/jama.2015.10945. PMID 26393848
- [Background] Wolff M, Sundquist K, Larsson Lonn S, Midlov P. Impact of yoga on blood pressure and quality of life in patients with hypertension - a controlled trial in primary care, matched for systolic blood pressure. BMC Cardiovasc Disord. 2013 Dec 7;13:111. doi: 10.1186/1471-2261-13-111. PMID 24314119
- [Background] Vickers AJ, Altman DG. Statistics notes: Analysing controlled trials with baseline and follow up measurements. BMJ. 2001 Nov 10;323(7321):1123-4. doi: 10.1136/bmj.323.7321.1123. No abstract available. PMID 11701584
- See also: Council MR. Developing and evaluating complex interventions: new guidance 2008 — http://www.mrc.ac.uk/complexinterventionsguidance